CLINICAL TRIAL: NCT02572726
Title: Integration of Neuroimaging and Transcranial Magnetic Stimulation: an Exploration of the Neuroplasticity of Endogenous Analgesia in Health and Chronic Pain
Brief Title: An Exploration of the Neuroplasticity of Endogenous Analgesia in Health and Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 0106-15_CTIL
Record Dates: First submitted 2015-10-06; First posted 2015-10-09 (Estimated); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- active rTMS (Active Comparator): active repeated transcranial magnetic stimulation over primary motor cortex along 5-10 daily sessions
  Interventions: Device: active repeated transcranial magnetic stimulation
- 'sham' rTMS (Sham Comparator): 'sham' repeated transcranial magnetic stimulation over primary motor cortex along 5-10 daily sessions
  Interventions: Device: 'sham' repeated transcranial magnetic stimulation

INTERVENTIONS:
Device: active repeated transcranial magnetic stimulation — ten daily sessions with active 10Hz 20 min-long stimulation over the primary motor cortex
  Arms: active rTMS
Device: 'sham' repeated transcranial magnetic stimulation — ten daily sessions with 'sham' 10Hz 20 min-long stimulation over the primary motor cortex
  Arms: 'sham' rTMS

SUMMARY:
Transcranial magnetic stimulation (TMS) is a neurophysiological tool for studying cortical functions, and in addition, has an analgesic therapeutic effect whose underlying mechanism is unknown. The proposed research will use TMS in conjunction with brain imaging and electrophysiology to examine cortical plasticity and connectivity modifications induced by repetitive TMS (rTMS) targeted to affect cortical regions associated with endogenous analgesia (EA). This will be carried out in both healthy and chronic pain (fibromyalgia) states. rTMS analgesic intervention, targeted to the motor cortex (M1) will be preceded and followed by structural and functional magnetic resonance imaging (fMRI), and Diffusion Tensor Imaging (DTI). This will be done in order to examine alterations of cortical and brainstem mechanisms involved in EA and to investigate connectivity changes between cortical and sub-cortical regions of the EA networks. The latter as well as EA efficiency and pain-related personality variables will be used to assess individual differences in neuroplasticity within the EA systems in both healthy subjects and chronic pain patients.

DETAILED DESCRIPTION:
Transcranial magnetic stimulation (TMS) is a neurophysiological tool for studying cortical functions, and in addition, has an analgesic therapeutic effect whose underlying mechanism is unknown. The proposed research will use TMS in conjunction with brain imaging and electrophysiology to examine cortical plasticity and connectivity modifications induced by repetitive TMS (rTMS) targeted to affect cortical regions associated with endogenous analgesia (EA). This will be carried out in both healthy and chronic pain (fibromyalgia) states. rTMS analgesic intervention, targeted to the motor cortex (M1) will be preceded and followed by structural and functional magnetic resonance imaging (fMRI), and Diffusion Tensor Imaging (DTI). This will be done in order to examine alterations of cortical and brainstem mechanisms involved in EA and to investigate connectivity changes between cortical and sub-cortical regions of the EA networks. The latter as well as EA efficiency and pain-related personality variables will be used to assess individual differences in neuroplasticity within the EA systems in both healthy subjects and chronic pain patients .

ELIGIBILITY:
Inclusion Criteria:

* a prior FMS diagnosis by a rheumatologist or pain specialist based on American College of Rheumatology (ACR) preliminary diagnostic criteria for fibromyalgia
* healthy subjects - no pain/psychiatry/neurological diseases

Exclusion Criteria:

* other chronic pain, psychiatric or neurological diseases. All will be asked to withdraw from any pain-relieving medications for 24h before the testing.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-10-11 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
rTMS-induced change in fibromyalgia pain level | through study completion, an average of 2 year
  Fibromyalgia pain level will be measured using the numerical pain scale; the patients will be asked to rate their mean pain level over the last 5 days

SECONDARY OUTCOMES:
treatment-induced changes of white-matter connectivity of the brain | through study completion, an average of 2 year
  White-matter connectivity will be measured using the method of diffusion tensor imaging of the brain

CONTACTS AND LOCATIONS:
Overall Officials: David Yarnitsky, MD, Prof, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel